CLINICAL TRIAL: NCT05317572
Title: Comparison of Three Different Doses of Intrathecal Morphine for Analgesia After Cesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Ilke Tamdogan, Physician, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CSITM2020
Record Dates: First submitted 2022-03-04; First posted 2022-04-08 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Cesarean Section; Spinal Anesthesia; Postoperative Analgesia
Keywords: Postoperative pain; Intrathecal morphine
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: The patients were randomly divided into three groups of 50patients each. In the system where computer generated random numbers (SPSS v23.0, IBM,- Page 2 of 6 [DRAFT] -NewYork, USA) were used,
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients were randomly divided into three groups of 50patients each. In the system where computer generated random numbers (SPSS v23.0, IBM,- Page 2 of 6 [DRAFT] -NewYork, USA) were used, groups were determined at a ratio of 1:1:1 . Sealed and sequentially numbered envelopes were created. One hour before the operation, an experienced anesthesiologist, who was not involved in the intraoperative and postoperative follow-up of the patient and would only perform the spinal anesthesia procedure, opened a sealed opaque sealed envelope to learn the group that the patient would be included in. There were two different physicians who performed intraoperative and postoperative follow-up. Both of the follow-up physicians were blind to the patient group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Active Comparator): Group 1: Spinal Anesthesia (10 mg hyperbaric bupivacaine + 20 mcg fentanyl+ 80 mcg intrathecal morphine) + iv Fentanyl-PCA
  Interventions: Drug: 80 mcg intrathecal morphine
- Group 2 (Active Comparator): Group 2: Spinal Anesthesia (10 mg hyperbaric bupivacaine + 20 mcg fentanyl+ 120 mcg intrathecal morphine) + iv Fentanyl-PCA
  Interventions: Drug: 120 mcg intrathecal morphine
- Group 3 (Active Comparator): Group 3: Spinal Anesthesia (10 mg hyperbaric bupivacaine + 20 mcg fentanyl+ 160 mcg intrathecal morphine) + iv Fentanyl-PCA
  Interventions: Drug: 160 mcg intrathecal morphine

INTERVENTIONS:
Drug: 80 mcg intrathecal morphine — İntraoperative Management:
  Spinal anesthesia was administered to each patient in a sitting position, after aseptic conditions were achieved with a midline approach. A 25 gauge pencil point spinal needle was placed in the L3-4 or L4-5 space. Upon aspiration of clear cerebrospinal fluid (CSF), 10 mg of hyperbaric bupivacaine, 20 mcg of fentanyl and 80 micrograms of morphine were injected into the intrathecal space together with the determined morphine doses.
  Postoperative analgesia management:
  Diclofenac sodium 2 × 75 mg was administered intramuscularly to all patients. All patients received iv Patient Controlled Analgesia (PCA) prepared with fentanyl postoperatively. For patients with pain VAS score of 5 or more, meperidine was administered at a rate of 25 mg each time and with a total daily dose of 200 mg.
  Arms: Group 1
Drug: 120 mcg intrathecal morphine — İntraoperative Management:
  Spinal anesthesia was administered to each patient in a sitting position, after aseptic conditions were achieved with a midline approach. A 25 gauge pencil point spinal needle was placed in the L3-4 or L4-5 space. Upon aspiration of clear cerebrospinal fluid (CSF), 10 mg of hyperbaric bupivacaine, 20 mcg of fentanyl and 120 micrograms of morphine were injected into the intrathecal space together with the determined morphine doses.
  Postoperative analgesia management:
  Diclofenac sodium 2 × 75 mg was administered intramuscularly to all patients. All patients received iv Patient Controlled Analgesia (PCA) prepared with fentanyl postoperatively. For patients with pain VAS score of 5 or more, meperidine was administered at a rate of 25 mg each time and with a total daily dose of 200 mg.
  Arms: Group 2
Drug: 160 mcg intrathecal morphine — İntraoperative Management:
  Spinal anesthesia was administered to each patient in a sitting position, after aseptic conditions were achieved with a midline approach. A 25 gauge pencil point spinal needle was placed in the L3-4 or L4-5 space. Upon aspiration of clear cerebrospinal fluid (CSF), 10 mg of hyperbaric bupivacaine, 20 mcg of fentanyl and 160 mcg of morphine were injected into the intrathecal space together with the determined morphine doses.
  Postoperative analgesia management:
  Diclofenac sodium 2 × 75 mg was administered intramuscularly to all patients. All patients received iv Patient Controlled Analgesia (PCA) prepared with fentanyl postoperatively. For patients with pain VAS score of 5 or more, meperidine was administered at a rate of 25 mg each time and with a total daily dose of 200 mg.
  Arms: Group 3

SUMMARY:
In our study, It was aimed to determine the dose of morphine that provides the most effective analgesia with the least incidence of side effects in the postoperative period.

DETAILED DESCRIPTION:
Spinal anesthesia is a widely used method in cesarean section operations. It has become a popular practice to add opioids to local anesthetic agents to improve the quality and prolong the duration of intraoperative and postoperative analgesia. Morphine and fentanyl are commonly used opioids for this purpose. In cesarean sections, intrathecal morphine (ITM) is preferred for postoperative analgesia due to its slow onset and long-term analgesia, and intrathecal fentanyl is preferred for intraoperative analgesia due to its faster onset of action.

ITM can cause side effects such as nausea, vomiting, itching, sedation and respiratory depression. The quality of analgesia and the incidence of side effects may vary depending on the ITM dose used. There are studies indicating that reducing the dose of ITM results in good quality, long-term analgesia with a low incidence of side effects. However, the ideal dose of ITM providing optimal postoperative analgesia with the lowest incidence of side effects for cesarean section has not been determined yet in the literature. For this purpose, in this study it was compared the postoperative analgesia efficiency and incidence of side effects of three different ITM doses in order to contribute to the literature.

Patients were divided into three groups:

Group 1: 10 mg hyperbaric bupivacaine + 20 mcg fentanyl+ 80 mcg intrathecal morphine was administered.

Group 2: 10 mg hyperbaric bupivacaine + 20 mcg fentanyl+ 120 mcg intrathecal morphine was administered.

Group 3: 10 mg hyperbaric bupivacaine + 20 mcg fentanyl+ 160 mcg intrathecal morphine was administered.

All patients received iv Patient Controlled Analgesia (PCA) prepared with fentanyl postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing cesarean section
* Between the ages of 18-40,
* ASA II,
* Pregnant women with gestational week > 36

Exclusion Criteria:

* Not accepting regional anesthesia,
* İnfection at the injection site,
* Coagulopathy, bleeding diathesis,
* Severe hypovolemia,
* İncrease in intracranial pressure,
* Pregnant women with problems such as severe aortic stenosis, severe mitral stenosis for which spinal anesthesia is contraindicated,
* Patients with a history of allergy to any drug included in the study protocol

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Fentanyl consumption in the first 24 hours after surgery | Postoperative Day 2
  Fentanyl consumption in the first 24 hours was measured. Patients were able to request opioids via a PCA device when their VAS score is above 4 at rest and during activity (coughing and walking).

SECONDARY OUTCOMES:
Post-operative acute pain | Postoperative Day 2
  Pain status at rest and while activity (coughing and walking) was assessed by VAS scores at 0, 8, 24, 30, and 48 hours after surgery. The VAS is an 11-point numeric scale which ranges from 0 to 10 at rest and during activity.
The incidences of post-operative nausea and vomiting (PONV) | Postoperative Day 2
  The severity of postoperative nausea and vomiting (PONV) was assessed using a Numeric rating scale(NRS) at 0, 8, 24, 30, and 48 hours after surgery. If a score of 3 or more is recorded, ondansetron 0,1 mg/kg iv was administered.
The incidence of side effects related to opioid use | Postoperative Day 2
  Complications related to opioid use such as pruritus, fatigue, sedation or respiratory depression was recorded
Bromage Score Comparison | Postoperative 2nd hour.
  After spinal anesthesia was administered, motor block was evaluated according to the Bromage scale. Bromage score and motor block removal times were noted at the intraoperative 5th, 30th minutes, at the end of the operation, at the postoperative 30th minute and at the 2nd hour.
APGAR score | The 5th minute APGAR score was recorded.
  The 5th minute APGAR score was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: ilke tamdoğan, Principal Investigator — Ondokuz Mayıs University Faculty of Medicine
Locations (1):
- Ondokuz Mayıs University Faculty of Medicine, Samsun, Turkey (Türkiye)

REFERENCES:
- [Result] Palmer CM, Emerson S, Volgoropolous D, Alves D. Dose-response relationship of intrathecal morphine for postcesarean analgesia. Anesthesiology. 1999 Feb;90(2):437-44. doi: 10.1097/00000542-199902000-00018. PMID 9952150
- [Result] Baraka A, Noueihid R, Hajj S. Intrathecal injection of morphine for obstetric analgesia. Anesthesiology. 1981 Feb;54(2):136-40. doi: 10.1097/00000542-198102000-00007. PMID 7008655
- [Result] Weigl W, Bierylo A, Wielgus M, Krzemien-Wiczynska S, Kolacz M, Dabrowski MJ. Perioperative analgesia after intrathecal fentanyl and morphine or morphine alone for cesarean section: A randomized controlled study. Medicine (Baltimore). 2017 Dec;96(48):e8892. doi: 10.1097/MD.0000000000008892. PMID 29310376
- [Result] Sarvela J, Halonen P, Soikkeli A, Korttila K. A double-blinded, randomized comparison of intrathecal and epidural morphine for elective cesarean delivery. Anesth Analg. 2002 Aug;95(2):436-40, table of contents. doi: 10.1097/00000539-200208000-00037. PMID 12145067